CLINICAL TRIAL: NCT05535387
Title: Integrated Smart Speaker/Mobile Application to Promote Positive Parenting Among Caregivers of Youth With Challenging Behaviors
Brief Title: Integrated Smart Speaker Promoting Positive Parenting Among Caregivers of Youth With Challenging Behaviors
Acronym: FamilyNet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MH124577
Record Dates: First submitted 2022-02-07; First posted 2022-09-10 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Oppositional Defiant Disorder; Conduct Disorder
MeSH Terms: conditions — Oppositional Defiant Disorder; Conduct Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FamilyNet smart speaker/mobile application (Experimental): In a 4-week period, families will use a prototype of the FamilyNet integrated and coordinated smart speaker/mobile application designed to provide families with in-situ experiential support for building positive behavior plans.
  Interventions: Behavioral: FamilyNet smart speaker/mobile application

INTERVENTIONS:
Behavioral: FamilyNet smart speaker/mobile application — In a 4-week period, families will use a prototype of the FamilyNet integrated and coordinated smart speaker/mobile application designed to provide families with in-situ experiential support for building positive behavior plans. The prototype FamilyNet program will guide families in creating and implementing positive behavior plans to foster positive child behavior, consistent parenting, and promote a positive parent-child relationship.

SUMMARY:
This project will develop and evaluate the feasibility of an integrated smart speaker and mobile/web-based application, "FamilyNet" (FN) to assist parents in implementing empirically supported behavioral parenting strategies to promote positive behavior change in their children. The FamilyNet system will help parents to create a positively framed, individualized behavioral plan for their child(ren), and then provide prompts, reminders, and tracking tools to help them effectively implement that plan. Once developed, FamilyNet will be field tested for usability and usefulness with a group of parents who have children ages 10-17 years exhibiting challenging behaviors. Establishing feasibility of this innovative parenting tool will have important implications for harnessing smart speaker and mobile/web technologies to provide parents in-situ support with parenting challenges; parents' effective implementation of empirically supported parenting strategies is likely to increase children's prosocial behaviors and reduce problematic behaviors, thus reducing their risk for long-term behavioral problems.

DETAILED DESCRIPTION:
This project will develop and establish feasibility of an integrated smart speaker and mobile/web application, FamilyNet, designed to help parents utilize best practices in behavioral parent training to create and implement personalized behavior plans for their children. The FamilyNet system will integrate mobile app, smart speaker technology, and website technologies to assist families in creating their behavior plan, and then will track compliance, timelines, incentives, and other details to assist parents in following through and maintaining the behavior change program that they have created. After development, the intervention program will be pilot-tested with up to 35 families of youth ages 10-17 with challenging behaviors.

Primary parents will complete measures of parenting practices and child behavior prior to using the FamilyNet system, and again after having access to the program for 4 weeks. During the intervention period, user information will be tracked. Post-intervention measures will also include primary parents' perceptions of usability and acceptability of and satisfaction with the FamilyNet system. Children will also complete satisfaction questionnaires at the post- intervention assessment. Data will be analyzed to determine the degree to which families are able to utilize the FamilyNet interface and report finding it helpful.

ELIGIBILITY:
Inclusion criteria:

1. Primary parent/caregiver who has a child ages 10- to 17-years-old who lives with them at least half the time
2. Has a smartphone and access to email
3. Speaks English

Exclusion criteria:

a. The target-age child has a developmental disability severe enough that the child is unable to speak and/or follow simple directions.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire 11-17 - Emotional Problems Subscale | Baseline (T1), 4 weeks after baseline (T2)
  Strengths and Difficulties Questionnaire 4-17 (SDQ; Goodman, 1997) is used to measure the child's overall adjustment. The SDQ is a brief, valid, reliable, and commonly used parent-report questionnaire about child behavior. The instrument includes 25 items that assess child challenging behaviors (emotional symptoms, conduct problems, hyperactivity/inattention), peer relationships, and prosocial behavior, with 5 items measuring each subscale. Respondents answer on a 3-point scale from 0 to 2 (0 = "Not true;" 2 = "Certainly true"). For the Emotional Problems Subscale, scores for the 5 items are summed together; the subscale score can range from 0 to 10. Higher scores indicate worse adjustment (worse outcome).
Strengths and Difficulties Questionnaire 11-17 - Conduct Problems Subscale | Baseline (T1), 4 weeks after baseline (T2)
  Strengths and Difficulties Questionnaire 4-17 (SDQ; Goodman, 1997) is used to measure the child's overall adjustment. The SDQ is a brief, valid, reliable, and commonly used parent-report questionnaire about child behavior. The instrument includes 25 items that assess child challenging behaviors (emotional symptoms, conduct problems, hyperactivity/inattention), peer relationships, and prosocial behavior, with 5 items measuring each subscale. Respondents answer on a 3-point scale from 0 to 2 (0 = "Not true;" 2 = "Certainly true"). For the Conduct Problems Subscale, scores for the 5 items are summed together; the subscale score can range from 0 to 10. Higher scores indicate worse adjustment (worse outcome).
Strengths and Difficulties Questionnaire 11-17 - Hyperactivity Subscale | Time Frame: Baseline (T1), 4 weeks after baseline (T2)
  Strengths and Difficulties Questionnaire 4-17 (SDQ; Goodman, 1997) is used to measure the child's overall adjustment. The SDQ is a brief, valid, reliable, and commonly used parent-report questionnaire about child behavior. The instrument includes 25 items that assess child challenging behaviors (emotional symptoms, conduct problems, hyperactivity/inattention), peer relationships, and prosocial behavior, with 5 items measuring each subscale. Respondents answer on a 3-point scale from 0 to 2 (0 = "Not true;" 2 = "Certainly true"). For the Hyperactivity Subscale, scores for the 5 items are summed together; the subscale score can range from 0 to 10. Higher scores indicate worse adjustment (worse outcome).
Strengths and Difficulties Questionnaire 11-17 - Peer Problems Subscale | Baseline (T1), 4 weeks after baseline (T2)
  Strengths and Difficulties Questionnaire 4-17 (SDQ; Goodman, 1997) is used to measure the child's overall adjustment. The SDQ is a brief, valid, reliable, and commonly used parent-report questionnaire about child behavior. The instrument includes 25 items that assess child challenging behaviors (emotional symptoms, conduct problems, hyperactivity/inattention), peer relationships, and prosocial behavior, with 5 items measuring each subscale. Respondents answer on a 3-point scale from 0 to 2 (0 = "Not true;" 2 = "Certainly true"). For the Peer Problems Subscale, scores for the 5 items are summed together; the subscale score can range from 0 to 10. Higher scores indicate worse adjustment (worse outcome).
Strengths and Difficulties Questionnaire 11-17 - Prosocial Subscale | Baseline (T1), 4 weeks after baseline (T2)
  Strengths and Difficulties Questionnaire 4-17 (SDQ; Goodman, 1997) is used to measure the child's overall adjustment. The SDQ is a brief, valid, reliable, and commonly used parent-report questionnaire about child behavior. The instrument includes 25 items that assess child challenging behaviors (emotional symptoms, conduct problems, hyperactivity/inattention), peer relationships, and prosocial behavior, with 5 items measuring each subscale. Respondents answer on a 3-point scale from 0 to 2 (0 = "Not true;" 2 = "Certainly true"). For the Prosocial Subscale, scores for the 5 items are summed together; the subscale score can range from 0 to 10. Higher scores indicate better adjustment (better outcome).
Strengths and Difficulties Questionnaire 11-17 - Total Difficulties Score | Baseline (T1), 4 weeks after baseline (T2)
  Strengths and Difficulties Questionnaire 4-17 (SDQ; Goodman, 1997) is used to measure the child's overall adjustment. The SDQ is a brief, valid, reliable, and commonly used parent-report questionnaire about child behavior. The instrument includes 25 items that assess child challenging behaviors (emotional symptoms, conduct problems, hyperactivity/inattention), peer relationships, and prosocial behavior, with 5 items measuring each subscale. Respondents answer on a 3-point scale from 0 to 2 (0 = "Not true;" 2 = "Certainly true"). For the Total Difficulties Score, subscale scores for the Emotional Problems, Conduct Problems, Hyperactivity, and Peer Problems items are summed together; the Total Difficulties score can range from 0 to 40. Higher scores indicate worse adjustment (worse outcome).
Program Acceptability - Parent Perception of Improvement | At 4 weeks after baseline (T2)
  Measure Description: Parents' perceptions of improvement in their child's behavior was measured with 4 items of the Program Acceptability - Parent Perception of Improvement Subscale measure at T2, 4 weeks after baseline. Parents indicate their perceptions of recent change in their child's positive behavior and their relationship with their child. Respondents answer items on a 5-point scale (e.g. 1 = Considerably worse; 5 = Greatly improved). Scores on these 4 items are averaged together; subscale scores range from 1 to 5. Higher scores indicate parent perceptions of more improvement (better outcome).
Program Acceptability - Parent Satisfaction Subscale - Parent Report | At 4 weeks after baseline (T2)
  Parent Satisfaction was measured with 10 items of the Program Acceptability - Parent Satisfaction Subscale measure at T2, 4 weeks after baseline, asking the extent to which parents found that the FamilyNet program was helpful, enjoyable, addressed important issues, helped them follow through on their behavior change plan, helped them manage their child's behavior more effectively, was the type of help they wanted, and their overall satisfaction with the program. Respondents answer items on a 7-point scale (e.g. 1 = Not at all; 7 = Very much). Scores on these 10 items are averaged together; subscale scores range from 1 to 7. Higher scores indicate better parent satisfaction.
Program Acceptability - Child Satisfaction Subscale - Child Report | At 4 weeks after baseline (T2)
  Child Satisfaction was measured with 5 items of the Program Acceptability - Child Satisfaction Subscale measure at post-treatment, asking the extent to which the child found that the FamilyNet program was helpful and enjoyable, and their overall satisfaction with the program. Respondents answer items on a 7-point scale (e.g. 1 = Not at all; 7 = Very much). Scores on these 5 items are averaged together; subscale scores range from 1 to 7. Higher scores indicate better child satisfaction.
System Usability Scale - Parent Report | At 4 weeks after baseline (T2)
  Parents' perceptions of the usability of the FamilyNet program is measured with the System Usability Scale (SUS), a commonly used 10-item scale that measures subjective perceptions of usability. Items are answered on a 5-point scale (0=Strongly disagree; 4=Strongly agree); scores on the scale are summed and multiplied by 2.5, such that they range from 0 to 100, with higher scores indicating better usability. The SUS has been normed, and scoring produces an overall usability "grade" (Brooke, 1996; Sauro, 2011). This measure is obtained from the parents at post-test.
System Usability Scale - Child Report | At 4 weeks after baseline (T2)
  Child perceptions of the usability of the FamilyNet program is measured with the System Usability Scale (SUS), a commonly used 10-item scale that measures subjective perceptions of usability. Items are answered on a 5-point scale (0=Strongly disagree; 4=Strongly agree); scores on the scale are summed and multiplied by 2.5, such that they range from 0 to 100, with higher scores indicating better usability (better outcome). The SUS has been normed, and scoring produces an overall usability "grade" (Brooke, 1996; Sauro, 2011). This measure is obtained from the youth at post-test.

SECONDARY OUTCOMES:
Parenting Practices Inventory - Inconsistent Discipline Subscale | Baseline (T1), 4 weeks after baseline (T2)
  The Parenting Practices Inventory (PPI) - Inconsistent Discipline Subscale (Metzler, Taylor, & Foster, 2006) was used to measure the degree to which the parents are inconsistent in their discipline practices. Parents answer 4 items about inconsistent discipline practices on a 7-point frequency scale (1 = Never; 7 = Always). Scores on these 4 items are averaged together; the subscale scores range from 1 to 7. Higher scores indicate more inconsistent discipline practices (worse outcome).
Parenting Practices Inventory - Positive Reinforcement Subscale | Baseline (T1), 4 weeks after baseline (T2)
  The Parenting Practices Inventory (PPI) - Positive Reinforcement Subscale (Metzler, Taylor, & Foster, 2006) was used to measure how much parents utilize positive reinforcement to promote positive behavior in their children. Parents answer 6 items about their likelihood of using different positive reinforcement techniques when their child behaves well or does a good job, on a 7-point scale (1 = Not at all likely; 7 = Extremely likely), 1 item about how often in an average week they praise or reward their child for doing a good job at home or school, on a 7-point scale (1 = Less than once per week; 7 = More than 10 times per day), and 2 items about how many times they have used positive reinforcement in the past 2 days for anything their child did well, on a 7-point scale (1 = Never; 7 = More than 7 times). Scores on these 9 items are averaged together; the Positive Reinforcement subscale scores range from 1 to 7. Higher scores indicate more positive reinforcement (better outcome).
CASY Child-Parent Relationship Scales - Parent-Child Conflict subscale | Baseline (T1), 4 weeks after baseline (T2)
  The CASY Parent-Child Relationship Scales - Parent-Child Conflict Subscale (Metzler, Biglan, Ary, & Li, 1998) is used to measure conflict between the parent and child. Items were originally adapted from Prinz, Foster, Kent, & O'Leary (1979). For the Parent-Child Conflict Subscale, 4 items ask parents how often four different conflict situations happened over the past week; parents answer on a 7-point frequency scale (1= Never; 7 = more than 7 times). Scores on these 4 items are averaged together; subscale scores range from 1 to 7. Higher scores indicate more parent-child conflict (worse outcome).
CASY Child-Parent Relationship Scales - Positive Family Relations Subscale | Baseline (T1), 4 weeks after baseline (T2)
  The CASY Parent-Child Relationship Scales - Positive Family Relations Subscale (Metzler, Biglan, Ary, & Li, 1998) is used to measure positive relationships between the parent and child. Items were originally adapted from Moos and Moos (1986). For the Positive Family Relations Subscale, 6 items ask parents about the degree to which they have had a positive relationship with their child (3 items) and in the family in general (3 items) over the past month; parents answer on a 7-point "how true" scale (1= Never true; 7 = Always true). Scores on these 6 items are averaged together; subscale scores range from 1 to 7. Higher scores indicate a more positive relationship (better outcome).
Program-Targeted Parenting Practices - Frequency Subscale | Baseline (T1), 4 weeks after baseline (T2)
  The frequency of parents' engagement in the parenting practices targeted by the FamilyNet intervention is measured via the Program-Targeted Parenting Practices - Frequency Subscale (Metzler, Smith, Feil, & Marquez, 2023). Created for this study, these 8 items ask parents to report the frequency with which they have engaged in target parenting practices in the past 4 weeks; parents report their frequency on a 6-point scale (0 = "Never in the past month;" 5 = "Every day"). Averaged scores range from 0 to 5, with higher scores indicating more frequent parental engagement in the target activities (better outcome).
Program-Targeted Parenting Practices - Parental Self-Efficacy Subscale | Baseline (T1), 4 weeks after baseline (T2)
  Parents' self-efficacy for engaging in the parenting practices targeted by the FamilyNet intervention is measured via the Program-Targeted Parenting Practices - Parental Self-Efficacy Subscale (Metzler, Smith, Feil, & Marquez, 2023). Created for this study, these 6 items ask parents to rate how confident they are that they know how to do a series of parenting practices targeted by the program, on a scale of 1 to 10 (1 = Not confident at all; 10 = Highly confident). Averaged scores range from 1 to 10, with higher scores indicating greater parental self-efficacy in doing the targeted behavior (better outcome).
Parent Daily Report of Child Behavior, Positive Behavior Subscale | Baseline (T1), 4 weeks after baseline (T2)
  The Parent Daily Report (PDR; Chamberlain & Reid, 1987) is used to measure parents' report of their children's positive and negative behaviors over the past 24 hours. For the PDR Positive Behavior Subscale, parents are asked to indicate the extent to which 7 positive behaviors occurred in the past 24 hours on a 4-point scale (0 = Not at all; 3 = A lot). The scores from these 7 items are averaged together, and the average score ranges from 0 to 3. Higher scores indicate more positive behavior (better outcome).
Parent Daily Report of Child Behavior, Negative Behavior Subscale | Baseline (T1), 4 weeks after baseline (T2)
  The Parent Daily Report (PDR; Chamberlain & Reid, 1987) is used to measure parents' report of their children's positive and negative behaviors over the past 24 hours. For the PDR Negative Behavior Subscale, parents are asked to indicate the extent to which 19 negative behaviors occurred in the past 24 hours on a 7-point scale (0 = 0; 6 = 6 or more). The scores from these 19 items are averaged together, and the average score ranges from 0 to 6. Higher scores indicate more negative behavior (worse outcome).
Families' Usage of the FamilyNet Program - Number of Families that Used the Program | At 4 weeks after baseline (T2)
  Families' usage of the FamilyNet program is measured through usage metrics collected on the back-end database, including the number of families that used the program and the number of times the program was used by families. For the Number of Families that Used the Program metric, families are identified either as (a) used the program at least once, or (b) did not use the program at all. "Usage" is defined as either the parent or the child used the program at least once during the program period (after the initial monitoring period). Higher levels for all usage metrics indicate greater program use.
Families' Usage of the FamilyNet Program - Number of Times the Program was Used | At 4 weeks after baseline (T2)
  Families' usage of the FamilyNet program is measured through usage metrics collected on the back-end database, including the number of families that used the program and the number of times the program was used by families. For number of Times the Program was Used, each instance of a family's "usage," defined as either the parent or the child using the program, was counted over the course of the intervention period (after the initial monitoring period). Higher levels for all usage metrics indicate greater program use.

CONTACTS AND LOCATIONS:
Overall Officials: David R. Smith, PhD, Principal Investigator — Oregon Research Behavioral Intervention Strategies, Inc.
Locations (1):
- Oregon Research Behavioral Intervention Strategies, Inc., Springfield, Oregon, United States

REFERENCES:
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Background] Brooke, J. (1996). SUS-A quick and dirty usability scale. In P. W. Jordan, B. Thomas, B. A. Weerdmeester, & I. L. McClelland (Eds.), Usability evaluation in industry (Vol. 189, pp. 169-194). London, UK: Taylor & Francis.
- [Background] Sauro, J. (2011). A practical guide to the system usability scale: Background, benchmarks & best practices. Denver, CO: Measuring Usability LLC.
- [Background] Metzler, C.W., Taylor, T.K., & Foster, E.M. (2006). Associations between specific parental discipline practices and specific dimensions of young children's behavior problems. Unpublished technical report.
- [Background] Metzler, C. W., Biglan, A., Ary, D. V., & Li, F. (1998). The stability and validity of early adolescents' reports of parenting constructs. Journal of Family Psychology, 12(4), 600-619.
- [Background] Prinz RJ, Foster S, Kent RN, O'Leary KD. Multivariate assessment of conflict in distressed and nondistressed mother-adolescent dyads. J Appl Behav Anal. 1979 Winter;12(4):691-700. doi: 10.1901/jaba.1979.12-691. PMID 541311
- [Background] Moos, R. H., & Moos, B. A. (1986). Manual for the Family Environment Scale. Palo Alto, CA: Consulting Psychologists Press.
- [Background] Chamberlain, P., & Reid, J. B. (1987). Parent observation and report of child symptoms. Behavioral Assessment, 9(1), 97-109.